CLINICAL TRIAL: NCT00763542
Title: A Randomized Controlled Trial Comparing (1) a Combined Treatment of CBT for Substance Use Disorders (SUD) and Trauma-focused Structured Writing Therapy With (2) CBT for SUD Alone in Patients With Comorbid SUD and PTSD
Brief Title: Combined Treatment for Patients With Comorbid Substance Use Disorders and Post-traumatic Stress Disorder (PTSD): an Integration of Cognitive-behavioral Treatment (CBT) and Trauma-focused Structured Writing Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Proffesor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-KP-342
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Substance-Related Disorders; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Combined treatment: CBT for SUD plus structured writing therapy for PTSD
  Interventions: Behavioral: CBT for SUD; Behavioral: Structured writing therapy for PTSD
- II (Active Comparator): CBT for SUD only
  Interventions: Behavioral: CBT for SUD

INTERVENTIONS:
Behavioral: CBT for SUD — CBT for SUD focuses on patient-motivation, self-control strategies and relapse-prevention.
Behavioral: Structured writing therapy for PTSD — Patients progress through three stages, in which instructions for writing and feedback by therapists are successively aimed at achieving trauma processing, cognitive restructuring and social sharing of a traumatic event.
  Arms: I

SUMMARY:
This study is a randomized controlled trial comparing two treatments for patients with comorbid substance use disorder (SUD) and post-traumatic stress disorder (PTSD) conducted within two different routine clinical settings for the treatment of SUD, namely (a) a day-care and inpatient setting and (b) an outpatient setting. Participants will be randomly assigned to either (1) a combination of cognitive-behavioral treatment (CBT) for SUD and trauma-focused structured writing therapy, or (2) CBT for SUD alone. Randomization will take place separately for each setting. It is expected that the combined treatment is significantly more effective in reducing symptoms of SUD as well as PTSD than CBT for SUD alone. Outcome measures will be assessed at pre-treatment, post-treatment as well as 3 months, 6 months and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of substance abuse or substance dependence according to DSM-IV
* Diagnosis of PTSD according to the DSM-IV or subthreshold PTSD (at least one re-experiencing symptom plus either three avoidance/numbing or two hyperarousal symptoms are present)
* 18 years or older
* Sufficient fluency in Dutch or English to complete treatment and research procedures

Exclusion Criteria:

* Severe psychiatric problems that may interfere with study participation or that require more intensive clinical care than can be offered in the present study (e.g., dementia, psychotic symptoms, depression with suicidal ideation, manic episode and borderline personality disorder)
* Receiving concurrent psychotherapy
* Participants using tranquilizers are required to terminate medication use before inclusion
* Participants using anti-depressant medication are required to stabilize medication use before inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Substance use assessed with the Time-Line Follow-Back Interview (TLFB; Sobell & Sobell, 1996) | Pre-treatment, Post-treatment; 3 months follow-up; 6 months; 12 months follow-up
PTSD symptom severity assessed with the Posttraumatic Diagnostic Scale (PDS; Foa et al., 1997) | Pre-treatment, Post-treatment, 3 months follow-up, 6 months; 12 months follow-up
DSM-IV diagnoses of SUD and PTSD assessed with the Structured Clinical Interview for the DSM-IV (SCID) | Pre-treatment, Post-treatment, 3 months follow-up, 6 months; 12 months follow-up

SECONDARY OUTCOMES:
Inventory of Drug Use Consequences (INDUC-2r) | Pre-treatment, Post-treatment, 3 months follow-up, 6 months; 12 months follow-up
Trauma-related appraisals assessed with the Posttraumatic Cognitions Inventory (PTCI) | Pre-treatment, Post-treatment, 3 months, 6 months, 12 months follow-up
Response to intrusions assessed with the Response to Intrusions Questionnaire (RIQ) | Pre-treatment, Post-treatment, 3 months, 6 months, 12 months follow-up
Metacognitions concerning alcohol and/or drug-use assessed with the Positive Alcohol Metacognitions Scale (PAMS) | Pre-treatment, Post-treatment, 3 months, 6 months, 12 months follow-up
Difficulties in Emotion regulation (DERS) | Pre-treatment, Post-treatment, 3-months, 6 months; 12 months follow-up
Interpretation of PTSD-symptoms (PTSD-IPSI) | Pre-treatment, Post-treatment, 3 months; 6 months, 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul MG Emmelkamp, Professor, Principal Investigator — University of Amsterdam; Debora van Dam, MSc, Study Director — University of Amsterdam; Ellen Vedel, PhD, Study Chair — JellinekMentrum; Thomas Ehring, PhD, Study Chair — University of Amsterdam
Locations (1):
- JellinekMentrum, Amsterdam, Netherlands